CLINICAL TRIAL: NCT00503958
Title: Liverpool Lung Project
Brief Title: Liverpool Lung Project: Risk Factors and Genetic Markers in Healthy Participants and Patients With Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Liverpool Cancer Research Centre (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: ULCRC-LLP; CDR0000554297 (Registry Identifier: PDQ (Physician Data Query)); EU-20735
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2007-11

CONDITIONS: Health Status Unknown; Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer; health status unknown
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — DNA Methylation; Gene Expression Profiling; Epidemiologic Studies; Biopsy

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: DNA stability analysis
Genetic: gene expression analysis
Other: epidemiologic study
Other: study of socioeconomic and demographic variables
Procedure: biopsy
Procedure: evaluation of cancer risk factors
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Environmental exposure and genetic predisposition may affect the risk of developing cancer later in life. Learning about genetic markers and the long-term effects of environmental exposure may help the study of lung cancer in the future.

PURPOSE: This research study is looking at risk factors and genetic markers in healthy participants and in patients with lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To prepare a molecular genetic and epidemiological risk assessment model based on the analysis of environmental exposures and genetic predisposition, which will provide an algorithm to measure an individual's risk for developing lung cancer.
* To develop an archive of specimens relating to at-risk individuals and those with lung cancer.
* To redefine lung cancer based on molecular pathology using the fields of expression and methylation profiling, and genetic instability.
* To identify and assess novel markers of pre-carcinogenesis in our high-risk populations.
* To facilitate the development of new intervention strategies (i.e., chemoprevention).

OUTLINE: This is a multicenter study.

Participants and/or patients undergo tumor tissue, sputum, and blood sample collection periodically. Samples are analyzed via fields of expression and methylation profiling and genetic instability. Samples are also archived.

Complete lifetime lifestyle, residential, environmental tobacco smoke, and occupational history are assessed in the first year and then in year five and year ten. Participants who return for follow-up complete a shorter questionnaire aimed at recording change over the interval since their last attendance.

PROJECTED ACCRUAL: 800 patients and 7,500 healthy participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Prospective cohort:

  * All residents (n=326,000), aged 45-79, within the designated Liverpool postcode study area will be eligible for entry into the study

    * 7,500 people will be randomly selected from this population via general practitioner's (GP's) lists held by each Primary Care Trust
    * All the GP's who have practices within the study area will be asked to collaborate with the project
* Case-control:

  * Patients: Newly diagnosed cases of primary lung cancer

    * All cases of epithelial tumors of the trachea, bronchus, and lung will be included
  * Two controls per case who are matched for age (+/- 2 years) and gender and will be randomly selected from the Liverpool Lung Project prospective cohort

PATIENT CHARACTERISTICS:

* Inclusion Criteria:

  * Prospective cohort:

    * Age 45-79
    * Living within the Liverpool electoral wards
  * Case-control:

    * Upper age limit of 80 years old
    * Resident within Liverpool Lung Project area
* Exclusion Criteria:

  * Both cohorts:

    * Unable to provide competent informed consent
    * Ineligible to approach based on consultant/clinical team advice
    * Infectious respiratory disease (i.e., chest infection and are on antibiotics) within the past 3 months
    * Untreated pulmonary tuberculosis within the past 3 months

PRIOR CONCURRENT THERAPY:

* Participant and/or patient must not have had any of the following treatments within the last 3 months and is not planning to undergo any of them:

  * Cardiac surgery
  * Thoracic surgery
  * Carotid artery surgery
  * Abdominal surgery
  * Chemotherapy
  * Deep x-ray therapy

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8300 (Estimated)
Dates: Start 1998-08

PRIMARY OUTCOMES:
Prepare a molecular genetic and epidemiological risk assessment model based on the analysis of environmental exposures and genetic predisposition, which will provide an algorithm to measure an individual's risk for developing lung cancer
Develop an archive of specimens relating to at-risk individuals and those with lung cancer
Redefine lung cancer based on molecular pathology using the fields of expression and methylation profiling, and genetic instability
Identify and assess novel markers of pre-carcinogenesis in high-risk populations
Facilitate the development of new intervention strategies (i.e., chemoprevention)

CONTACTS AND LOCATIONS:
Overall Officials: John K. Field, MA, BDS, PhD, FRCPath, Principal Investigator — University of Liverpool Cancer Research Centre
Locations (5):
- United Kingdom (5):
  - University of Liverpool Cancer Research Centre, Liverpool, England
  - Aintree University Hospital, Liverpool, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - Whiston Hospital, Prescot Merseyside, England
  - Cardiothoracic Centre - Liverpool, Liverpool

REFERENCES:
- [Background] Field JK, Smith DL, Duffy S, Cassidy A. The Liverpool Lung Project research protocol. Int J Oncol. 2005 Dec;27(6):1633-45. PMID 16273220